CLINICAL TRIAL: NCT04121572
Title: EtCO2 for Monitoring and Predicting Severity of DKA in Pediatric Emergency, Doha, Qatar.
Status: Recruiting | Type: Observational
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Principal Investigator, DR. KHALID AL-ANSARI, Director of Pediatric Emergency Center's, Hamad Medical Corporation
Other Study IDs: MRC-01-17-103
Record Dates: First submitted 2019-10-08; First posted 2019-10-10 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Diabetes Mellitus
Keywords: Diabetic ketoacidosis; End tidal carbon dioxide; Capnography
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Ketoacidosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Nasal cannula capnography — Capnography: a continuous wave form of the CO2 level with the digital reading of CO2 level at end of expiration

SUMMARY:
Metabolic acidosis is one of the important and life-threatening pathophysiological changes in DKA and its monitoring is essential. It is known that the level of carbon dioxide (CO2) in the blood is correlating with the degree of metabolic acidosis. The CO2 level can be measured via the exhaled air by nasal cannula capnography (EtCO2) which is currently utilized to monitor the patient ventilation in many situations. Our primary objective is to study the degree of correlation between continuous EtCO2 monitoring and the severity of metabolic acidosis in blood gas measurement in patients with diabetic keto-acidosis (DKA). Secondary objectives are: ability of EtCO2 in ruling in or out DKA; discriminating the different severity grades of DKA. It is a cross-sectional, observational, prospective cohort study in convenience sample of children presenting with clinical manifestations consistent with DKA. Will be conducted in pediatric Emergency Center, Hamad General Hospital. Will include all DKA patients and excluding any condition or medication that affect the acid-base status.

DETAILED DESCRIPTION:
The study will be conducted in pediatric emergency center, Hamad General Hospital, a recognized academic institution, in Doha, Qatar.

The DKA was defined as: hyperglycemia (blood glucose >11 mmol/L or 200 mg/dL), venous pH <7.3 and/ or bicarbonate <15 mmol/L, and the association with, ketonemia, and ketonuria. The severity of DKA is categorized as mild (venous pH <7.3 or bicarbonate <15 mmol/L), moderate (venous pH <7.2 or bicarbonate < 10 mmol/L) and severe (venous pH < 7.1 or bicarbonate <5 mmol/L).

Eligible patients are all children with already known or newly diagnosed diabetics, regardless weather has been enrolled in previous encounter or not.

The patients with the following criteria are excluded: older than 14 years of age, airway obstruction, chest infection, complex congenital heart disease, Congestive heart failure, central or peripheral neurological disorders, hyper/hypothermia, and sever pain.

Physicians and nurses, and research assistance staff will be trained in the use of nasal capnography including the proper size, connection and wave forms shapes and its interpretation.

ELIGIBILITY:
Inclusion Criteria:

All children with already known or newly diagnosed diabetics, regardless weather has been enrolled in previous encounter or not.

Exclusion Criteria:

1. Older than 14 years of age
2. Airway obstruction
3. Chest infection
4. Complex congenital heart disease
5. Congestive heart failure
6. Central or peripheral neurological disorders
7. Hyper/hypothermia
8. Severe pain

Max Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: known or newly diagnosed diabetics children between the age group of 0- 14 years
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-10-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
To utilize capnography as a noninvasive tool for the detection and monitoring of DKA | 2 years
  Capnography measures exhaled CO2 which is an indicator of the presence and severity of metabolic acidosis caused by DKA.

SECONDARY OUTCOMES:
To find the ability of EtCO2 in ruling in or out DKA | 2 years
  by correlating the of exhaled CO2 level to the level of Bicarbonate level in blood sample we can assess if the patient is having DKA on arrival or had it and get out of it during the management

OTHER OUTCOMES:
To evaluate the different severity grades of DKA using EtCO2 Monitoring | 2years
  by correlating the severity of DKA based on the bicarbonate level to the exhaled CO2 level

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Khalid Alansari, Principal Investigator — Hamad Medical Corporation
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: Undecided